CLINICAL TRIAL: NCT05322135
Title: A Pilot Study of Glutamine PET Imaging of Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0739; NCI-2022-02415 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2022-03-15; First posted 2022-04-11 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — 4-(3-fluoropropyl)glutamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET scan (Experimental): PET scans: an 11C-Glutamine PET scan and an 18F-FSPG PET scan. A small tube (called an IV) will be placed in a vein in your arm through which you will receive the radioactive material for the PET scan(s).
  Interventions: Drug: 18F-FSPG; Drug: 11C-Glutamine

INTERVENTIONS:
Drug: 18F-FSPG — Given by vein (IV)
Drug: 11C-Glutamine — Given by vein (IV)

SUMMARY:
We propose a focused, prospective pilot clinical imaging trial to evaluate 11C-Gln PET/CT followed by 18F-FSPG PET/CT in 20 HNSCC patients. Imaging metrics that are common to PET (e.g. SUVmax, peak or mean) will be determined.

This study will also allow the acquisition of additional safety and biodistribution data, as, to date, only a limited number of patients have been evaluated with 11C-Gln as a direct PET imaging biomarker of Gln uptake. To date, no adverse side effects have been observed. We do not anticipate any toxicity since this tracer is a naturally-occurring essential amino acid in high abundance and is administered at sub-pharmacologic doses.

A long-term goal of these preliminary studies is to validate the utility of Gln PET imaging metrics for HNSCC and to expand this imaging technique to additional patients in prospective cohorts of patients with HNSCC.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this trial is to evaluate the ability of 11C-Gln and 18F-FSPG PET imaging to detect tumors in patients with HNSCC.

Hypotheses: 11C-Gln PET and 18F-FSPG PET will yield standardized uptake values SUVs; within HNSCC primary and metastatic lesions that are significantly higher relative to SUV of background tissue.

Primary Outcome Measures

11C-Gln standardized uptake value (SUV) including SUVmax, SUVpeak, and SUVmean for tumors and normal tissue 18F-FSPG standardized uptake value (SUV) including SUVmax, SUVpeak, and SUVmean for tumors and normal tissue

Secondary Objectives:

A secondary objective of this trial is to compare PET imaging data to standard-of-care MRI or CT. Another secondary objective is to determine the tumor-to-background ratios (TBR) for 11C-Gln and 18F-FSPG. A third secondary objective is to determine the safety of 11C-Gln.

Hypotheses: 11C-Gln PET and 18F-FSPG PET will detect additional sites of disease that are not visualized by CT or MRI. In addition, tumor-to-background ratios (TBR) for either tracer will exceed 2. Finally, 11C-Gln will be safe at the doses administered in this study.

Secondary Outcome Measures:

Number of lesions. Lesion count will be determined on a per patient basis. Tumor size (e.g., long-axis diameter, short-axis diameter, tumor volume) derived from standard-of-care (SOC) CT or MRI. Tumor size will be defined according to RECIST v1.1 [10] with the longest diameter measured for tumor lesions and the short-axis diameter measured for malignant lymph nodes.

Tumor-to-background ratios (TBR) for 11C-Gln and 18F-FSPG Adverse events associated with 11C-Gln

Exploratory Objectives:

An exploratory objective of this trial is to compare 11C-Gln PET/CT and 18F-FSPG PET/CT imaging to conventional 18F-FDG PET when feasible. Another exploratory objective is to compare uptake of 11C-Gln and 18F-FSPG between HPV-positive and HPV-negative patients.

Hypothesis: The SUVmax and TBR for 11C-Gln PET or 18F-FSPG PET will be greater than 18F-FDG PET. We also hypothesize based on the published expression data that 11C-Gln and 18F-FSPG avidity will differ between HPV-positive and negative patients, with 11C-Gln having higher uptake in HPV-positive patients, while 18F-FSPG will have higher uptake in HPV-negative patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. Pathologically or cytologically confirmed diagnosis of head and neck squamous cell carcinoma (HNSCC);
3. Documented results from (or scheduled to undergo) CT or MRI as a SOC procedure within 42 days prior to baseline investigational 11C-Gln PET/CT and 18F-FSPG PET/CT;
4. Measurable disease by RECIST v1.1 defined as tumor lesions with a longest diameter ≥ 10 mm and/or malignant lymph nodes with a short axis diameter ≥ 15 mm.
5. Ability to provide written informed consent in accordance with institutional policies.
6. Non-English speaking subject will be included. Verbal Translation Preparative Sheet (VTPS) short form will be utilized in consent non-English speaking subject

Exclusion Criteria:

1. Body weight ≥400 pounds or body habitus or disability that will not permit the imaging protocol to be performed;
2. Pregnant or lactating females.
3. Have an allergy to intravenous contrast
4. eGFR<30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
To establish the ability of 11C-Gln PET imaging to detect tumors in patients with (HNSCC) Head and Neck Squamous Cell Carcinoma NSCC. | through study completion, an average of 1 year
To establish the ability of the 18F-FSPG PET imaging to detect tumors in patients with (HNSCC) Head and Neck Squamous Cell Carcinoma NSCC. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Flynt, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT05322135/ICF_000.pdf